CLINICAL TRIAL: NCT03074071
Title: Enhancing Hope Among Patients With Poor-Prognosis Breast Cancer and Oncologists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TASMC-17-OG-0619-CTIL
Record Dates: First submitted 2017-02-23; First posted 2017-03-08 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Despair Among Cancer Patients and Oncologists
Keywords: Disambiguation, Depression, Burnout
MeSH Terms: conditions — Depression; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Subjects will be offered participation in workshops where techniques are taught for enhancing hopefulness. Validated questionnaires will be administered before and after this intervention to assess efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast Cancer patient (Active Comparator): Patients with Stage IV breast cancer will be taught to build hope by defining attainable goals for themselves in a Hope Enhancement Workshop.
  Interventions: Behavioral: Hope Enhancement Workshop
- Oncologists (Active Comparator): Oncologists will will be taught to build hope by defining attainable goals for themselves and for their patients in a Hope Enhancement Workshop.
  Interventions: Behavioral: Hope Enhancement Workshop

INTERVENTIONS:
Behavioral: Hope Enhancement Workshop — Participants in the workshops will be prompted and guided through exercises that help them get in touch with goals that are not explicitly related to cure of disease. These goals will include symptom relief and other personal and or professional objectives.

SUMMARY:
The study will access whether breast cancer patients and oncologists can become more hopeful after participating in a "hope enhancement workshop." Several validated tools, Adult Hope Scale (AHS), Herth Hope Index (HHI), Maslach Burnout Inventory (MBI)" and other quality of life parameter surveys, will be administered at specified intervals.

DETAILED DESCRIPTION:
The aim of the proposed research is to study the impact of hope interventions on the coping behavior of women with advanced breast cancer and physicians who provide care to patients with cancer.

It is the investigator's contention, that improved hopefulness among cancer patients can be manifest in improved Quality of Life (QOL). The challenge is to find specific interventions that can optimize hopefulness and thereby direct individuals to adopt behavior styles that contribute to a positive effect on QOL.

Two separate single-day interventions and hope applications will be developed for patients and oncologists, respectively. What will be common for each workshop is that there will be an experienced counselor designated as "coordinator" who will be in charge of implementing the program and monitoring group dynamics. The interventions will be structured with the program advancing from the identification of goals to the development of directions reasonable pathways for achieving the delineated goals. In addition to goal-directed exercises, the workshop will employ narrative techniques which utilize literary triggers as a springboard for reflective writing.

The smartphone-based application will prompt study participants on a daily basis to engage in additional, short activities designed to augment hopefulness, assess progress in achieving goals, and identifying challenges. In addition, the application will allow sustained interaction of workshop participants through social media exchange.

Course materials will be sent to study participants one week prior to the conduct of the workshop.

Baseline assessment of hopefulness will be carried out via the aforementioned validated scales on the day of the workshop.

Re-assessment of hopefulness will occur at the end of the day and at the 3- month interval visits.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (patient component of study)

* Diagnosis of invasive breast cancer that is Stage IV.
* Female, 18 years of age or older.
* Able to proficiently speak, read, write English.
* ECOG performance status between 0 and 3.
* Subjects must have a smartphone with at least "3rd generation" mobile technology, and willingness to download and utilize specialized application
* Expected to continue cancer care at the institution where cancer was begun for the duration of the study.

Inclusion Criteria (physician component of study)

* Board certification or board eligibility in any of the 3 oncologic disciplines:

  * Medical Oncology
  * Surgical Oncology
  * Radiation Oncology
* Able to proficiently speak, read, write English.
* Subjects must have a smartphone with at least "3rd generation" mobile technology, and willingness to download and utilize specialized application
* NB: There will not be active recruitment of physicians who are subordinate to the respective investigators. In the event that such a physician desires to enroll on the study, formal application will be made to the institutional ethics committees to verify that coercion has not taken place.

Exclusion Criteria:

Exclusion Criteria (applies to both patients and physicians)

* Participant actively undergoing psychotherapy for depression.
* Documented history of Alzheimer's disease or other forms of dementia.
* Participants practicing mindfulness meditation for an average of more than 1 hour/week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of the change in Hope Enhancement | The primary measurement will be carried out prior to and 3 months following the workshop
  Enhancement of hopefulness as measured by Adult Hope Scale
Measurement of the change in Hopefulness | The primary measurement will be carried out prior to and 3 months following the workshop
  Enhancement of hopefulness as measured by Herth Hope Index.
Measurement of the change in Quality of Life and Emotional Stress Anxiety | The primary measurement will be carried out prior to and 3 months following the workshop
  The study will measure QOL and emotional stress anxiety prior to and 3 months following the intervention. Towards these ends, we will use the Patient-Reported Outcomes Measurement Information System (PROMIS) scale (10-point version).
Measurement of the change in Quality of Life and Well Being | The primary measurement will be carried out prior to and 3 months following the workshop
  The study will measure QOL and well-being prior to and 3 months following the intervention. Towards these ends, we will use the Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being (FACIT-Sp-12) scale.

SECONDARY OUTCOMES:
Measurement of the change in burnout among oncologists | The measurement will be carried out prior to and 3 months following the workshop.
  The study will measure burnout among oncologists using the Maslach Burnout Inventory Scale (MBI) to gauge the willingness of oncologists to incorporate hope enhancement techniques to their clinical routine with patients following the workshop intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No